CLINICAL TRIAL: NCT02233023
Title: Matched Pair, Assessor Blinded, Open Label Clinical Trial to Assess the Ophthalmologic Safety of Long Term Oral Treatment With Pramipexole Compared to Bromocriptine or Other Dopamine Agonists in Patients With Parkinson's Disease
Brief Title: Ophthalmologic Safety of Long Term Treatment With Pramipexole Compared to Bromocriptine or Other Dopamine Agonists in Patients With Parkinson's Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 248.342
Record Dates: First submitted 2014-09-04; First posted 2014-09-08 (Estimated); Last update posted 2014-09-08 (Estimated); Status verified 2014-09

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Pramipexole; Bromocriptine

ARMS (2):
- Pramixpexole (Experimental)
  Interventions: Drug: Pramipexole
- Bromocriptine and other dopamine agonists (Active Comparator)
  Interventions: Drug: Bromocriptine and other dopamine agonists

INTERVENTIONS:
Drug: Pramipexole
  Arms: Pramixpexole
Drug: Bromocriptine and other dopamine agonists
  Arms: Bromocriptine and other dopamine agonists

SUMMARY:
Study to assess and compare the safety of long term oral treatment for Parkinson's Disease with pramipexole versus bromocriptine or other dopamine agonists, by measuring cross-sectional the incidence of ophthalmologic disturbances, especially signs of retinal degeneration, in a matched pair design

ELIGIBILITY:
Inclusion Criteria:

* Patients with idiopathic Parkinson's Disease
* Patients treated consecutively with either pramipexole or bromocriptine (or other dopamine agonists except ropinirole) for at least two and a half years (i.e. 30 months). Interruptions of ongoing dopamine agonists treatment for less than one month per year duration are acceptable, however, interruptions within the last 6 months are not acceptable. Patients currently participating in ongoing open-label extension trials with pramipexole may be included if they meet the requirement of 30 month treatment
* Written informed consent in accordance with Good Clinical Practice (GCP) and local legislation

Exclusion Criteria:

* Patients who have been treated less than two and a half years (i.e. 30 months) with their actual dopamine agonist (regardless of the duration of treatment with a previous dopamine agonist)
* Patient treated with ropinirole
* Patients with any of the following:

  * Patients with a hereditary retinal disease and/or a family history of hereditary retinal disease
  * Patients with a history of drug-induced retinopathies
  * Patients with a history of surgically or laser-treated diabetic retinopathy
* Patients with atypical parkinsonian syndromes due to drugs, metabolic disorders, encephalitis or degenerative diseases (e.g. progressive, supranuclear palsy, multisystem atrophy)
* Dementia or other disorders that could impair the signing of informed consent
* Patients who are participating in other drug studies or who receive other investigational drugs within 30 days prior to the first visit (patients currently participating in ongoing open-label extension trials with pramipexole may be included if they meet the requirement of 30 months treatment duration

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 705 (Actual)
Dates: Start 1998-06; Primary Completion 2000-06 (Actual)

PRIMARY OUTCOMES:
Incidence of drug related signs of retinal degeneration | up to 8 months
  based on the evaluation of assessors blind to the treatment allocation

SECONDARY OUTCOMES:
Assessment of ophthalmological history | within 2 month after neurologic visit
Assessment of visual acuity | within 2 month after neurologic visit
Number of abnormal findings in clinical examination in miosis and mydriasis | within 2 month after neurologic visit
  including ophthalmoscopy
Assessment of intraocular pressure (mmHg) | within 2 month after neurologic visit
Assessment of colour vision | within 2 month after neurologic visit
  using the Hardy-Rand-Rittler (H-R-R) pseudoisochromatic plates
Findings in kinetic perimetry | within 2 month after neurologic visit
Percentage of patients with elevated dark adaptation thresholds | within 2 month after neurologic visit
Assessment of Parkinson's Disease stage rated by modified Hoehn and Yahr Scale | within less than 2 months before ophthalmologic visit
Assessment of Parkinson's Disease stage rated of unified Parkinson's Disease Rating Scale (UPDRS) Part IV | within less than 2 months before ophthalmologic visit
Number of patients with adverse events | up to 2 month after neurologic visit
Findings in standardised electroretinography (ERG) | within 2 monhts after neurologic visit
  performed according to International Standardization Committee for the Electrophysiology of Vision (ISCEV) standard